CLINICAL TRIAL: NCT05932784
Title: The Impact of Aortic Valve Compression During Cardio-pulmonary Resuscitation on Patients With Out-of-hospital Cardiac Arrest: A Single-center Observational Study Using Transesophageal Echocardiography
Brief Title: The Impact of Aortic Valve Compression During Cardio-pulmonary Resuscitation on Patients With Out-of-hospital Cardiac Arrest
Acronym: AVC in OHCA
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 109070-F-2
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHCA patients receiving TEE: Out-of-hospital cardiac arrest (OHCA) patients undergo transesophageal echocardiography (TEE) during resuscitation to determine if their aortic valve is being compressed.
  Interventions: Device: transesophageal echocardiography

INTERVENTIONS:
Device: transesophageal echocardiography — Utilizing transesophageal echocardiography (TEE) during resuscitation allows medical professionals to determine if a patient's aortic valve is being compressed while receiving chest compressions, providing valuable insight to optimize the resuscitation process.
  Other Names: TEE

SUMMARY:
Purpose:

This study aims to find out if the current way of performing chest compressions during resuscitation for patients who have suffered a cardiac arrest outside of the hospital is affecting their chances of recovery. Recent research suggests that more than half of these patients receive chest compressions near their aortic valve, which might block blood flow and make their condition worse. We will use a special imaging technique called transesophageal echocardiography (TEE) during resuscitation to see if compressions near the aortic valve impact patient outcomes.

Methods:

We will conduct a study with patients who have suffered a cardiac arrest outside of the hospital and are receiving TEE during resuscitation in the emergency department. Some patients will not be included in the study, such as those who recover quickly before the TEE is done, those who need other treatments before they recover, those with an unclear compression site, or those with poor or missing TEE images. We will divide the patients into two groups: those with compressions near their aortic valve and those without. We will collect information on the patients, the TEE recordings, the resuscitation process, and important time points. We will mainly look at whether the patients recover and maintain a steady heartbeat. We will also examine other factors like their carbon dioxide levels, whether they recover at all, if they survive to be admitted to the hospital, if they survive to be discharged, and if they have good brain function when they leave the hospital. We plan to have 37 patients in each group for accurate results.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 20 or older who arrived at the ED with non-traumatic OHCA and underwent TEE during resuscitation

Exclusion Criteria:

1. Early ROSC before obtaining TEE image;
2. Insert the REBOA before ROSC;
3. Initiate ECMO flow before ROSC;
4. Cannot identify compression site on TEE;
5. Poor quality of TEE image;
6. Missing TEE image.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20 or older who arrived at the ED with non-traumatic OHCA and underwent TEE during resuscitation were enrolled, except for those meeting the following exclusion criteria: 1) Early ROSC before obtaining TEE image; 2) Insertion of REBOA before ROSC; 3) Initiation of ECMO flow before ROSC; 4) Unidentifiable compression site on TEE; 5) Poor quality TEE image; 6) Missing TEE image
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
sustained return of spontaneous circulation (ROSC) | 20 minutes after ROSC
  successful restoration and maintenance of a patient's heartbeat and blood circulation after undergoing cardiopulmonary resuscitation (CPR) for at least 20 minutes

SECONDARY OUTCOMES:
Any return of spontaneous circulation (ROSC) | 1 minutes after ROSC
survival to admission | 48 hours after ROSC
survival to discharge | 6 months after ROSC
discharge with favorable neurological outcomes | 6 months after ROSC
end-tidal carbon dioxide (EtCO2) | During resuscitation

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No